CLINICAL TRIAL: NCT01840579
Title: A Phase I Study of MK-3475 Alone in Subjects With Advanced Solid Tumors and in Combination With Platinum-Doublet Chemotherapy or Immunotherapy in Subjects With Advanced Non-Small Cell Lung Cancer/Extensive-Disease Small Cell Lung Cancer.
Brief Title: Study of Pembrolizumab (MK-3475) Monotherapy in Advanced Solid Tumors and Pembrolizumab Combination Therapy in Advanced Non-small Cell Lung Cancer/ Extensive-disease Small Cell Lung Cancer (MK-3475-011/KEYNOTE-011)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3475-011; 132249 (Registry Identifier: JAPIC-CTI); MK-3475-011 (Other: Merck); KEYNOTE-011 (Other: Merck)
Record Dates: First submitted 2013-04-23; First posted 2013-04-25 (Estimated); Results first posted 2021-03-22 (Actual); Last update posted 2021-06-22 (Actual); Status verified 2021-05

CONDITIONS: Solid Tumor; Non-small Cell Lung Cancer; Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma | interventions — pembrolizumab; Cisplatin; Pemetrexed; Paclitaxel; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Ipilimumab; Etoposide; etoposide phosphate; Granulocyte Colony-Stimulating Factor; pegfilgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Pembrolizumab 2 mg/kg (Experimental): In Part A, participants receive intravenous (IV) Pembrolizumab 2 mg/kg on Day 1 of Cycle 1 (28 days), Cycle 2 and any additional cycles (14 days).
  Interventions: Biological: Pembrolizumab 2 mg/kg
- Pembrolizumab 10 mg/kg (Experimental): In Part A, participants receive IV Pembrolizumab 10 mg/kg on Day 1 of Cycle 1 (28 days), Cycle 2 and any additional cycles (14 days).
  Interventions: Biological: Pembrolizumab 10 mg/kg
- Pembrolizumab+Cisplatin/Pemetrexed (Experimental): In Part B, participants receive IV Pembrolizumab 200 mg + IV Cisplatin 75 mg/m^2 + IV Pemetrexed 500 mg/m^2 on Day 1 of each 21-day cycle for a maximum of 4 cycles. After completion of the initial therapy, maintenance therapy with IV pemetrexed in combination with IV pembrolizumab is permitted per standard of care, followed by IV pembrolizumab 200 mg every 3 weeks.
  Interventions: Biological: Pembrolizumab 200 mg; Drug: Cisplatin 75 mg/m^2; Drug: Pemetrexed 500 mg/m^2
- Pembrolizumab+Carboplatin/Pemetrexed (Experimental): In Part B, participants receive IV Pembrolizumab 200 mg + IV Carboplatin Area Under The Curve (AUC) 5 mg/mL/minute + IV Pemetrexed 500 mg/m^2 on Day 1 of each 21-day cycle for a maximum of 4 cycles. After completion of the initial therapy, maintenance therapy with IV pemetrexed in combination with IV pembrolizumab is permitted per standard of care, followed by IV pembrolizumab 200 mg every 3 weeks.
  Interventions: Biological: Pembrolizumab 200 mg; Drug: Pemetrexed 500 mg/m^2; Drug: Carboplatin AUC 5 mg/mL/min
- Pembrolizumab+Carboplatin/Paclitaxel (Experimental): In Part C, participants receive IV Pembrolizumab 200 mg + IV Carboplatin AUC 6 mg/mL/minute + IV Paclitaxel 200 mg/m^2 on Day 1 of each 21-day cycle for a maximum of 4 cycles. After completion of the initial therapy, maintenance therapy with IV pembrolizumab 200 mg every 3 weeks.
  Interventions: Biological: Pembrolizumab 200 mg; Drug: Carboplatin AUC 6 mg/mL/min; Drug: Paclitaxel 200 mg/m^2
- Pembrolizumab+Carboplatin/Nab-paclitaxel (Experimental): In Part C, participants receive IV Pembrolizumab 200 mg + IV Carboplatin AUC 6 mg/mL/minute on Day 1 of each 21-day cycle + IV Nab-paclitaxel 100 mg/m^2 on Days 1, 8, and 15 of each 21-day cycle for a maximum of 4 cycles. After completion of the initial therapy, maintenance therapy with IV pembrolizumab 200 mg every 3 weeks.
  Interventions: Biological: Pembrolizumab 200 mg; Drug: Carboplatin AUC 6 mg/mL/min; Drug: Nab-paclitaxel 100 mg/m^2
- Pembrolizumab+Ipilimumab (Experimental): In Part D, participants receive IV Pembrolizumab 200 mg on Day 1 of each 21-day cycle + IV Ipilimumab 1 mg/kg on Day 1 of every other 21-day cycle (every 42 days) for a maximum of 18 cycles of Ipilimumab (35 doses of Pembrolizumab).
  Interventions: Biological: Pembrolizumab 200 mg; Biological: Ipilimumab 1 mg/kg
- Pembrolizumab+Cisplatin/Etoposide (Experimental): In Part E, participants receive IV Pembrolizumab 200 mg + IV Cisplatin 75 mg/m^2 on Day 1 of each 21-day cycle + IV Etoposide 100 mg/m^2 on Days 1, 2, and 3 of each 21-day cycle for a maximum of 4 cycles. After completion of the initial therapy, maintenance therapy with IV pembrolizumab 200 mg every 3 weeks.
  Interventions: Biological: Pembrolizumab 200 mg; Drug: Cisplatin 75 mg/m^2; Drug: Etoposide 100 mg/m^2
- Pembrolizumab+Carboplatin/Etoposide (Experimental): In Part E, participants receive IV Pembrolizumab 200 mg + IV Carboplatin AUC 5 mg/mL/minute on Day 1 of each 21-day cycle + IV Etoposide 100 mg/m^2 on Days 1, 2, and 3 of each 21-day cycle for a maximum of 4 cycles. After completion of the initial therapy, maintenance therapy with IV pembrolizumab 200 mg every 3 weeks.
  Interventions: Biological: Pembrolizumab 200 mg; Drug: Carboplatin AUC 5 mg/mL/min; Drug: Etoposide 100 mg/m^2
- Pembrolizumab+Cisplatin/Etoposide+G-CSF (Experimental): In Part E, participants receive IV Pembrolizumab 200 mg + IV Cisplatin 75 mg/m^2 on Day 1 of each 21-day cycle + IV Etoposide 100 mg/m^2 on Days 1, 2, and 3 of each 21-day cycle for a maximum of 4 cycles + lasting granulocyte colony-stimulating factor (G-CSF) (pegfilgrastim) 3.6 mg on Day 4 of Cycle 1. After completion of the initial therapy, maintenance therapy with IV pembrolizumab 200 mg every 3 weeks.
  Interventions: Biological: Pembrolizumab 200 mg; Drug: Cisplatin 75 mg/m^2; Drug: G-CSF (pegfilgrastim) 3.6 mg

INTERVENTIONS:
Biological: Pembrolizumab 2 mg/kg — Administered as an intravenous (IV) infusion on Day 1 of Cycle 1 (28 days), Cycle 2 (14 days), and Cycle 3 (14 days)
  Other Names: KEYTRUDA®
  Arms: Pembrolizumab 2 mg/kg
Biological: Pembrolizumab 10 mg/kg — Administered as an IV infusion on Day 1 of Cycle 1 (28 days), Cycle 2 (14 days), and Cycle 3 (14 days)
  Other Names: KEYTRUDA®
  Arms: Pembrolizumab 10 mg/kg
Biological: Pembrolizumab 200 mg — Administered as an IV infusion on Day 1 of each 21-day cycle
  Other Names: KEYTRUDA®
  Arms: Pembrolizumab+Carboplatin/Etoposide; Pembrolizumab+Carboplatin/Nab-paclitaxel; Pembrolizumab+Carboplatin/Paclitaxel; Pembrolizumab+Carboplatin/Pemetrexed; Pembrolizumab+Cisplatin/Etoposide; Pembrolizumab+Cisplatin/Etoposide+G-CSF; Pembrolizumab+Cisplatin/Pemetrexed; Pembrolizumab+Ipilimumab
Drug: Cisplatin 75 mg/m^2 — Administered as an IV infusion on Day 1 of each 21-day cycle
  Arms: Pembrolizumab+Cisplatin/Etoposide; Pembrolizumab+Cisplatin/Etoposide+G-CSF; Pembrolizumab+Cisplatin/Pemetrexed
Drug: Pemetrexed 500 mg/m^2 — Administered as an IV infusion on Day 1 of each 21-day cycle
  Arms: Pembrolizumab+Carboplatin/Pemetrexed; Pembrolizumab+Cisplatin/Pemetrexed
Drug: Carboplatin AUC 5 mg/mL/min — Administered as an IV infusion on Day 1 of each 21-day cycle
  Arms: Pembrolizumab+Carboplatin/Etoposide; Pembrolizumab+Carboplatin/Pemetrexed
Drug: Carboplatin AUC 6 mg/mL/min — Administered as an IV infusion on Day 1 of each 21-day cycle
  Arms: Pembrolizumab+Carboplatin/Nab-paclitaxel; Pembrolizumab+Carboplatin/Paclitaxel
Drug: Paclitaxel 200 mg/m^2 — Administered as an IV infusion on Day 1 of each 21-day cycle
  Arms: Pembrolizumab+Carboplatin/Paclitaxel
Drug: Nab-paclitaxel 100 mg/m^2 — Administered as an IV infusion on Days 1, 8, and 15 of each 21-day cycle
  Other Names: ABRAXANE®
  Arms: Pembrolizumab+Carboplatin/Nab-paclitaxel
Biological: Ipilimumab 1 mg/kg — Administered as an IV infusion on Day 1 of every other 21-day cycle (every 42 days)
  Other Names: YERVOY®
  Arms: Pembrolizumab+Ipilimumab
Drug: Etoposide 100 mg/m^2 — Administered as an IV infusion on Days 1, 2, and 3 of each 21-day cycle
  Other Names: TOPOSAR®, VEPESID®, ETOPOPHOS®, EPOSIN®
  Arms: Pembrolizumab+Carboplatin/Etoposide; Pembrolizumab+Cisplatin/Etoposide
Drug: G-CSF (pegfilgrastim) 3.6 mg — Administered as a subcutaneous injection on Day 4 of Cycle 1
  Other Names: Neulasta®
  Arms: Pembrolizumab+Cisplatin/Etoposide+G-CSF

SUMMARY:
This study using pembrolizumab (MK-3475) will be done in 5 parts. In Part A, successive participant cohorts with advanced solid tumors will receive pembrolizumab to assess the safety and tolerability of monotherapy. In Parts B, C, and D, participants with advanced non-small cell lung cancer (NSCLC) will receive pembrolizumab in combination with either cisplatin/pemetrexed or carboplatin/pemetrexed (Part B); with either carboplatin/paclitaxel or carboplatin/nab-paclitaxel (Part C); or with ipilimumab (Part D) by non-random assignment to assess the safety and tolerability of the combination therapy. In Part E, participants with untreated Extensive-disease (ED) Small Cell Lung Cancer (SCLC) will receive pembrolizumab in combination with either cisplatin/etoposide, carboplatin/etoposide, or cisplatin/etoposide with prophylactic use of granulocyte colony-stimulating factor (lasting G-CSF [pegfilgrastim]) by non-random assignment to assess the safety and tolerability of the combination therapy.

ELIGIBILITY:
Inclusion Criteria:

* In Part A: has a histological or cytological diagnosis of solid tumor, progressive metastatic disease, or progressive locally advanced disease not amenable to local therapy
* In Part B, C, and D: has a histologically- or cytologically-confirmed diagnosis of NSCLC (Stage IIIB/IV) and are naïve to systemic therapy
* In Part C: has a histologically- or cytologically-confirmed diagnosis of squamous cancer
* In Part E: has a histologically- or cytologically-confirmed diagnosis of SCLC (ED stage) and are naïve to systemic therapy
* Has Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Has adequate organ function
* Female participants of reproductive potential must not be pregnant (negative urine or serum human chorionic gonadotropin test within 72 hours of study start)
* Female and male participants of reproductive potential must agree to use adequate contraception throughout the study period and for up to 120 days after the last dose of study therapy and for up to 180 days after the last dose of chemotherapeutic agents

Exclusion criteria:

* Has had cancer therapy within 2 weeks (Part E) or 4 weeks (Parts A, B, C, and D) prior to the first dose of study therapy, or not recovered from the adverse events of agents administered more than 4 weeks prior to the first dose of study therapy.

  * Part A: Chemotherapy, radiation therapy, biological therapy or kinase inhibitors
  * Parts B, C, D and E: Radiation therapy
* For Part B: has a histological diagnosis of squamous cancer
* Is currently participating or has participated in a study with an investigational agent or using an investigational device within 30 days of first dose of study therapy
* Is expected to require any other form of antineoplastic therapy while on study
* Is on chronic systemic steroid therapy within two weeks prior to the first dose of trial treatment or on any other form of immunosuppressive medication
* For Part C: Has pre-existing peripheral neuropathy that is ≥ Grade 2 by Common Terminology Criteria for Adverse Events version 4 criteria
* Has interstitial lung disease detected by chest computed tomography (CT), or a history of pneumonitis that required oral or intravenous glucocorticoids to assist with management. Lymphangitic spread of the NSCLC is not exclusionary.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2013-04-26 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Shimizu T, Seto T, Hirai F, Takenoyama M, Nosaki K, Tsurutani J, Kaneda H, Iwasa T, Kawakami H, Noguchi K, Shimamoto T, Nakagawa K. Phase 1 study of pembrolizumab (MK-3475; anti-PD-1 monoclonal antibody) in Japanese patients with advanced solid tumors. Invest New Drugs. 2016 Jun;34(3):347-54. doi: 10.1007/s10637-016-0347-6. Epub 2016 Mar 22. PMID 27000274
- [Derived] Nogami N, Umemura S, Kozuki T, Zenke Y, Ohtani J, Ishii M, Han S, Noguchi K, Horinouchi H. A phase 1 study of pembrolizumab plus ipilimumab as first-line treatment in Japanese patients with advanced non-small-cell lung cancer. Respir Investig. 2025 May;63(3):296-302. doi: 10.1016/j.resinv.2025.02.010. Epub 2025 Mar 3. PMID 40036983
- [Derived] Nogami N, Tokito T, Zenke Y, Satouchi M, Seto T, Saka H, Ohtani J, Han S, Noguchi K, Nishio M. Phase 1 study of pembrolizumab plus chemotherapy in Japanese patients with extensive-stage small-cell lung cancer. Invest New Drugs. 2024 Feb;42(1):136-144. doi: 10.1007/s10637-023-01411-1. Epub 2024 Feb 1. PMID 38300341
- [Derived] Kurata T, Nakagawa K, Satouchi M, Seto T, Sawada T, Han S, Homma M, Noguchi K, Nogami N. Phase 1 study of pembrolizumab plus chemotherapy as first-line treatment in Japanese patients with advanced NSCLC. Cancer Treat Res Commun. 2021;29:100458. doi: 10.1016/j.ctarc.2021.100458. Epub 2021 Sep 15. PMID 34607222
- See also: Merck Oncology Clinical Trials Information — http://merckoncologyclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Part A: Pembrolizumab 2 mg/kg: In Part A, participants received intravenous (IV) Pembrolizumab 2 mg/kg on Day 1 of Cycle 1 (28 days), Cycle 2 and any additional cycles (14 days).
- Part A: Pembrolizumab 10 mg/kg: In Part A, participants received IV Pembrolizumab 10 mg/kg on Day 1 of Cycle 1 (28 days), Cycle 2 and any additional cycles (14 days).
- Part B: Pembrolizumab+Cisplatin/Pemetrexed: In Part B, participants received IV Pembrolizumab 200 mg + IV Cisplatin 75 mg/m^2 + IV Pemetrexed 500 mg/m^2 on Day 1 of each 21-day cycle for a maximum of 4 cycles. After completion of the initial therapy, maintenance therapy with IV pemetrexed in combination with IV pembrolizumab is permitted per standard of care, followed by IV pembrolizumab 200 mg every 3 weeks.
- Part B: Pembrolizumab+Carboplatin/Pemetrexed: In Part B, participants receive IV Pembrolizumab 200 mg + IV Carboplatin Area Under The Curve (AUC) 5 mg/mL/minute + IV Pemetrexed 500 mg/m^2 on Day 1 of each 21-day cycle for a maximum of 4 cycles. After completion of the initial therapy, maintenance therapy with IV pemetrexed in combination with IV pembrolizumab is permitted per standard of care, followed by IV pembrolizumab 200 mg every 3 weeks.
- Part C: Pembrolizumab+Carboplatin/Paclitaxel: In Part C, participants received IV Pembrolizumab 200 mg + IV Carboplatin AUC 6 mg/mL/minute + IV Paclitaxel 200 mg/m^2 on Day 1 of each 21-day cycle for a maximum of 4 cycles. After completion of the initial therapy, maintenance therapy with IV pembrolizumab 200 mg every 3 weeks.
- Part C: Pembrolizumab+Carboplatin/Nabpaclitaxel: In Part C, participants received IV Pembrolizumab 200 mg + IV Carboplatin AUC 6 mg/mL/minute on Day 1 of each 21-day cycle + IV Nab-paclitaxel 100 mg/m^2 on Days 1, 8, and 15 of each 21-day cycle for a maximum of 4 cycles. After completion of the initial therapy, maintenance therapy with IV pembrolizumab 200 mg every 3 weeks.
- Part D: Pembrolizumab+Ipilimumab: In Part D, participants received IV Pembrolizumab 200 mg on Day 1 of each 21-day cycle + IV Ipilimumab 1 mg/kg on Day 1 of every other 21-day cycle (every 42 days) for a maximum of 18 cycles of Ipilimumab (35 doses of Pembrolizumab).
- Part E: Pembrolizumab+Cisplatin/Etoposide: In Part E, participants received IV Pembrolizumab 200 mg + IV Cisplatin 75 mg/m^2 on Day 1 of each 21-day cycle + IV Etoposide 100 mg/m^2 on Days 1, 2, and 3 of each 21-day cycle for a maximum of 4 cycles. After completion of the initial therapy, maintenance therapy with IV pembrolizumab 200 mg every 3 weeks.
- Part E: Pembrolizumab+Carboplatin/Etoposide: In Part E, participants received IV Pembrolizumab 200 mg + IV Carboplatin AUC 5 mg/mL/minute on Day 1 of each 21-day cycle + IV Etoposide 100 mg/m^2 on Days 1, 2, and 3 of each 21-day cycle for a maximum of 4 cycles. After completion of the initial therapy, maintenance therapy with IV pembrolizumab 200 mg every 3 weeks.
- Part E: Pembrolizumab+Cisplatin/Etoposide+G-CSF: In Part E, participants received IV Pembrolizumab 200 mg + IV Cisplatin 75 mg/m^2 on Day 1 of each 21-day cycle + IV Etoposide 100 mg/m^2 on Days 1, 2, and 3 of each 21-day cycle for a maximum of 4 cycles + lasting granulocyte colony-stimulating factor (G-CSF) (pegfilgrastim) 3.6 mg on Day 4 of Cycle 1. After completion of the initial therapy, maintenance therapy with IV pembrolizumab 200 mg every 3 weeks.
Period: Overall Study
Arm/Group | Part A: Pembrolizumab 2 mg/kg | Part A: Pembrolizumab 10 mg/kg | Part B: Pembrolizumab+Cisplatin/Pemetrexed | Part B: Pembrolizumab+Carboplatin/Pemetrexed | Part C: Pembrolizumab+Carboplatin/Paclitaxel | Part C: Pembrolizumab+Carboplatin/Nabpaclitaxel | Part D: Pembrolizumab+Ipilimumab | Part E: Pembrolizumab+Cisplatin/Etoposide | Part E: Pembrolizumab+Carboplatin/Etoposide | Part E: Pembrolizumab+Cisplatin/Etoposide+G-CSF
Started | 3 | 7 | 6 | 6 | 8 | 6 | 6 | 6 | 6 | 3
Completed | 0 | 0 | 4 | 3 | 4 | 2 | 4 | 3 | 3 | 0
Not Completed | 3 | 7 | 2 | 3 | 4 | 4 | 2 | 3 | 3 | 3
Not completed — Status not recorded | 0 | 0 | 2 | 3 | 4 | 3 | 0 | 3 | 3 | 3
Not completed — Progressive disease | 3 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Ongoing in study | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Follow-up ended by Sponsor | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A: Pembrolizumab 2 mg/kg | Part A: Pembrolizumab 10 mg/kg | Part B: Pembrolizumab+Cisplatin/Pemetrexed | Part B: Pembrolizumab+Carboplatin/Pemetrexed | Part C: Pembrolizumab+Carboplatin/Paclitaxel | Part C: Pembrolizumab+Carboplatin/Nabpaclitaxel | Part D: Pembrolizumab+Ipilimumab | Part E: Pembrolizumab+Cisplatin/Etoposide | Part E: Pembrolizumab+Carboplatin/Etoposide | Part E: Pembrolizumab+Cisplatin/Etoposide+G-CSF | Total
Number analyzed (Participants) | 3 | 7 | 6 | 6 | 8 | 6 | 6 | 6 | 6 | 3 | 57
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.3 (6.4) | 64.3 (13.6) | 57.3 (15.4) | 70.0 (6.0) | 66.6 (8.2) | 65.2 (11.8) | 66.0 (6.9) | 64.0 (3.6) | 64.7 (11.8) | 60.7 (8.1) | 64.4 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 1 | 1 | 0 | 0 | 0 | 3 | 2 | 2 | 14
  Male | 2 | 3 | 5 | 5 | 8 | 6 | 6 | 3 | 4 | 1 | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 7 | 6 | 6 | 8 | 6 | 6 | 6 | 6 | 3 | 57
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 3 | 7 | 6 | 6 | 8 | 6 | 6 | 6 | 6 | 3 | 57
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — An ECOG Performance Status of 0 (fully active, able to carry on all pre-disease performance without restriction) or 1 (restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature) was required for inclusion in the study. Participants were categorized by ECOG score.
  Participants
    ECOG = 0 | 2 | 2 | 3 | 2 | 1 | 1 | 0 | 2 | 2 | 3 | 18
    ECOG = 1 | 1 | 5 | 3 | 4 | 7 | 5 | 6 | 4 | 4 | 0 | 39

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced Dose-limiting Toxicities (DLTs)
Description: The following toxicities graded per the Common Terminology Criteria for Adverse Events version 4.0 (CTCAE v.4.0) were considered DLTs if judged by the investigator to be related to either study drug:
  * Grade (G) 4 neutropenia lasting >7 days
  * Grade 3 and Grade 4 febrile neutropenia
  * Grade 4 thrombocytopenia (<25,000/mm^3)
  * Grade 4 anemia
  * Grade 4 non-hematologic toxicity (not laboratory)
  * Grade 3 non-hematologic toxicity (not laboratory) lasting >3 days despite optimal supportive care
  * Any Grade 3 non-hematologic laboratory value if medical intervention is required to treat the participant or the abnormality persists for >7 days.
  * (Part D only) Missing the second dose of pembrolizumab (Cycle1 Day 22) due to drug-related adverse event
Time Frame: Cycle 1 (first dose and up to 4 weeks in Part A, 3 weeks in Parts B, C, E, and 6 weeks in Part D)
Population: The DLT analysis set included all participants who received at least at least 90% of the prescribed dose of pembrolizumab and the combination regimen and were evaluable for DLTs in the DLT evaluation period.
Measure: Count of Participants; unit: Participants
Groups:
- Part C: Pembrolizumab+Carboplatin/Nab-paclitaxel: In Part C, participants received IV Pembrolizumab 200 mg + IV Carboplatin AUC 6 mg/mL/minute on Day 1 of each 21-day cycle + IV Nab-paclitaxel 100 mg/m^2 on Days 1, 8, and 15 of each 21-day cycle for a maximum of 4 cycles. After completion of the initial therapy, maintenance therapy with IV pembrolizumab 200 mg every 3 weeks.
Arm/Group | Part A: Pembrolizumab 2 mg/kg | Part A: Pembrolizumab 10 mg/kg | Part B: Pembrolizumab+Cisplatin/Pemetrexed | Part B: Pembrolizumab+Carboplatin/Pemetrexed | Part C: Pembrolizumab+Carboplatin/Paclitaxel | Part C: Pembrolizumab+Carboplatin/Nab-paclitaxel | Part D: Pembrolizumab+Ipilimumab | Part E: Pembrolizumab+Cisplatin/Etoposide | Part E: Pembrolizumab+Carboplatin/Etoposide | Part E: Pembrolizumab+Cisplatin/Etoposide+G-CSF
Number analyzed (Participants) | 3 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 3
Participants | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 3 | 0 | 0

2. Primary Outcome: Number of Participants Who Experienced at Least One Adverse Event (AE)
Description: An adverse event is defined as any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An adverse event can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition that is temporally associated with the use of the Sponsor's product, is also an adverse event.
Time Frame: Up to approximately 51.3 months
Population: The analysis population consisted of all participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Pembrolizumab 2 mg/kg | Part A: Pembrolizumab 10 mg/kg | Part B: Pembrolizumab+Cisplatin/Pemetrexed | Part B: Pembrolizumab+Carboplatin/Pemetrexed | Part C: Pembrolizumab+Carboplatin/Paclitaxel | Part C: Pembrolizumab+Carboplatin/Nab-paclitaxel | Part D: Pembrolizumab+Ipilimumab | Part E: Pembrolizumab+Cisplatin/Etoposide | Part E: Pembrolizumab+Carboplatin/Etoposide | Part E: Pembrolizumab+Cisplatin/Etoposide+G-CSF
Number analyzed (Participants) | 3 | 7 | 6 | 6 | 8 | 6 | 6 | 6 | 6 | 3
Participants | 3 | 7 | 6 | 6 | 8 | 6 | 5 | 6 | 6 | 3

3. Primary Outcome: Number of Participants Who Discontinued Study Treatment Due to an Adverse Event (AE)
Description: as for outcome 2
Time Frame: Up to approximately 37.9 months
Population: The analysis population consisted of all participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Pembrolizumab 2 mg/kg | Part A: Pembrolizumab 10 mg/kg | Part B: Pembrolizumab+Cisplatin/Pemetrexed | Part B: Pembrolizumab+Carboplatin/Pemetrexed | Part C: Pembrolizumab+Carboplatin/Paclitaxel | Part C: Pembrolizumab+Carboplatin/Nab-paclitaxel | Part D: Pembrolizumab+Ipilimumab | Part E: Pembrolizumab+Cisplatin/Etoposide | Part E: Pembrolizumab+Carboplatin/Etoposide | Part E: Pembrolizumab+Cisplatin/Etoposide+G-CSF
Number analyzed (Participants) | 3 | 7 | 6 | 6 | 8 | 6 | 6 | 6 | 6 | 3
Participants | 0 | 0 | 1 | 5 | 4 | 3 | 2 | 1 | 1 | 0

4. Secondary Outcome: Maximum Serum Concentration (Cmax) of Pembrolizumab for Cycle 1: Parts A, B, C, D, and E
Description: Cmax was the maximum observed concentration of pembrolizumab in serum. For Part A, samples were collected on Day 1 at pre-dose, post-dose (to +30 min), 6 hour (hr) (±30 min), and 24hr; Days 2, 3, 8, 15, and 22 (±2 hr for Day 2 to Day 22) after completion of infusion. For Parts B, C, and E, samples were collected on Day 1 at pre-dose, post-dose (to +30 min), and 24hr; Day 5 (96hr was preferred, 72hr or 120hr were also acceptable, ±2 hr), and Day 15 (±24 hr) after completion of infusion. For Part D, samples were collected on Day 1 at pre-dose, post-dose (to +30 min), and 24hr; Day 5 (96hr was preferred, 72hr or 120hr were also acceptable, ±2 hr), Day 15, and Day 22 (±24 hr) after completion of infusion. Cycle 1 length for Part A was 28 days. Cycle 1 length for Parts B, C, and E was 21 days. Cycle 1 length for Part D was 42 days. Cmax is reported as geometric mean with a percent coefficient of variation. Per protocol, analysis for Cmax was planned for Parts A, B, C, D, and E.
Time Frame: At designated timepoints in Cycle 1 for Parts A, B, C, D, and E (up to approximately 22 days)
Population: The analysis population consisted of all participants who received pembrolizumab and contributed blood samples for analysis of Cmax in Parts A, B, C, D, and E Cycle 1.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Part A: Pembrolizumab 2 mg/kg | Part A: Pembrolizumab 10 mg/kg | Part B: Pembrolizumab+Cisplatin/Pemetrexed | Part B: Pembrolizumab+Carboplatin/Pemetrexed | Part C: Pembrolizumab+Carboplatin/Paclitaxel | Part C: Pembrolizumab+Carboplatin/Nab-paclitaxel | Part D: Pembrolizumab+Ipilimumab | Part E: Pembrolizumab+Cisplatin/Etoposide | Part E: Pembrolizumab+Carboplatin/Etoposide | Part E: Pembrolizumab+Cisplatin/Etoposide+G-CSF
Number analyzed (Participants) | 3 | 7 | 6 | 6 | 8 | 6 | 6 | 6 | 6 | 3
µg/mL | 47.4 (19) | 250 (23) | 52.51 (24.44) | 47.46 (17.04) | 56.39 (18.88) | 53.79 (14.18) | 72.71 (10.12) | 74.33 (14.04) | 84.55 (7.38) | 88.65 (19.14)

5. Secondary Outcome: Maximum Serum Concentration (Cmax) of Pembrolizumab for Cycle 2: Part A
Description: Cmax was the maximum observed concentration of pembrolizumab in serum. Blood sampling was taken for Part A on Day 1 of Cycle 2 at pre-dose and 0-30 minutes post-dose. Cycle 2 length for Part A was 14 days. Cmax is reported as geometric mean with a percent coefficient of variation (%CV). Per protocol, analysis for Cmax in Cycle 2 was only planned for Part A.
Time Frame: Cycle 2 Day 1 pre- and post-dose
Population: The analysis population consisted of all participants who received pembrolizumab and contributed blood samples for analysis of Cmax in Part A Cycle 2.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Part A: Pembrolizumab 2 mg/kg | Part A: Pembrolizumab 10 mg/kg
Number analyzed (Participants) | 3 | 6
µg/mL | 82.7 (12) | 322 (36)

6. Secondary Outcome: Maximum Serum Concentration (Cmax) of Pembrolizumab for Cycle 4: Parts A and D
Description: Cmax was the maximum observed concentration of pembrolizumab in serum. Blood sampling was taken for Part A on Day 1 of Cycle 4 at pre-dose and 0-30 minutes post-dose and for Part D on Day 22 of Cycle 4 at pre-dose (Day 1 of the following cycle prior to pembrolizumab infusion) and 0-30 minutes post-dose. Cycle 4 length for Part A was 14 days. Cycle 4 length for Part D was 42 days. Cmax is reported as geometric mean with a percent coefficient of variation (%CV). Per protocol, analysis for Cmax in Cycle 4 was only planned for Parts A and D.
Time Frame: Cycle 4 Day 1 pre- and post-dose (Part A) and Day 22 pre-dose (Day 1 of the following cycle prior to pembrolizumab infusion) and post-dose (Part D)
Population: The analysis population consisted of all participants who received pembrolizumab and contributed blood samples for analysis of Cmax in Cycle 4 Parts A and D.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Part A: Pembrolizumab 2 mg/kg | Part A: Pembrolizumab 10 mg/kg | Part D: Pembrolizumab+Ipilimumab
Number analyzed (Participants) | 2 | 3 | 3
µg/mL | 93.0 (44) | 367 (35) | 86.21 (3.59)

7. Secondary Outcome: Maximum Serum Concentration (Cmax) of Pembrolizumab for Cycle 6: Part A
Description: Cmax was the maximum observed concentration of pembrolizumab in serum. Blood sampling was taken for Part A on Day 1 of Cycle 6 at pre-dose and 0-30 minutes post-dose. Cycle 6 length for Part A was 14 days. Cmax is reported as geometric mean with a percent coefficient of variation (%CV). Per protocol, analysis for Cmax in Cycle 6 was only planned for Part A.
Time Frame: Cycle 6 Day 1 pre- and post-dose
Population: The analysis population consisted of all participants who received pembrolizumab and contributed blood samples for analysis of Cmax in Part A Cycle 6.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Part A: Pembrolizumab 2 mg/kg | Part A: Pembrolizumab 10 mg/kg
Number analyzed (Participants) | 2 | 2
µg/mL | 115 (15) | 286 (19)

8. Secondary Outcome: Maximum Serum Concentration (Cmax) of Pembrolizumab for Cycle 8: Parts A, B, C, and E
Description: Cmax was the maximum observed concentration of pembrolizumab in serum. Blood sampling was taken for Parts A, B, C and E on Day 1 of Cycle 8 at pre-dose and 0-30 minutes post-dose. Cycle 8 length for Part A was 14 days. Cycle 8 length for Parts B, C, and E was 21 days. Cmax is reported as geometric mean with a percent coefficient of variation (%CV). Per protocol, analysis for Cmax in Cycle 8 was only planned for Parts A, B, C, and E.
Time Frame: Cycle 8 Day 1 pre- and post-dose
Population: The analysis population consisted of all participants who received pembrolizumab and contributed blood samples for analysis of Cmax in Parts A, B, C, and E Cycle 8. There were no participants that contributed data for the analysis of Cmax for the Pembrolizumab+Cisplatin/Etoposide+G-CSF arm in Part E of Cycle 8.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Part A: Pembrolizumab 2 mg/kg | Part A: Pembrolizumab 10 mg/kg | Part B: Pembrolizumab+Cisplatin/Pemetrexed | Part B: Pembrolizumab+Carboplatin/Pemetrexed | Part C: Pembrolizumab+Carboplatin/Paclitaxel | Part C: Pembrolizumab+Carboplatin/Nab-paclitaxel | Part E: Pembrolizumab+Cisplatin/Etoposide | Part E: Pembrolizumab+Carboplatin/Etoposide | Part E: Pembrolizumab+Cisplatin/Etoposide+G-CSF
Number analyzed (Participants) | 2 | 1 | 2 | 3 | 1 | 2 | 1 | 3 | 0
µg/mL | 115 (15) | 298 (NA) — %CV was not planned to be calculated for ≤2 participants. | 124.47 (NA) — %CV was not planned to be calculated for ≤2 participants. | 95.51 (17.38) | 122.00 (NA) — %CV was not planned to be calculated for ≤2 participants. | 66.62 (NA) — %CV was not planned to be calculated for ≤2 participants. | 150.00 (NA) — %CV was not planned to be calculated for ≤2 participants. | 131.78 (9.46) |

9. Secondary Outcome: Maximum Serum Concentration (Cmax) of Pembrolizumab for Cycle 10: Part A
Description: Cmax was the maximum observed concentration of pembrolizumab in serum. Blood sampling was taken for Part A on Day 1 of Cycle 10 at pre-dose and 0-30 minutes post-dose. Cycle 10 length for Part A was 14 days. Cmax is reported as geometric mean with a percent coefficient of variation (%CV). Per protocol, analysis for Cmax in Cycle 10 was only planned for Part A.
Time Frame: Cycle 10 Day 1 pre- and post-dose
Population: The analysis population consisted of all participants who received pembrolizumab and contributed blood samples for analysis of Cmax in Part A Cycle 10.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Part A: Pembrolizumab 2 mg/kg | Part A: Pembrolizumab 10 mg/kg
Number analyzed (Participants) | 1 | 1
µg/mL | 133 (NA) — %CV was not planned to be calculated for ≤2 participants. | 266 (NA) — %CV was not planned to be calculated for ≤2 participants.

10. Secondary Outcome: Maximum Serum Concentration (Cmax) of Pembrolizumab for Cycle 12: Part A
Description: Cmax was the maximum observed concentration of pembrolizumab in serum. Blood sampling was taken for Part A on Day 1 of Cycle 12 at pre-dose and 0-30 minutes post-dose. Cycle 12 length for Part A was 14 days. Cmax is reported as geometric mean with a percent coefficient of variation (%CV). Per protocol, analysis for Cmax in Cycle 12 was only planned for Part A.
Time Frame: Cycle 12 Day 1 pre- and post-dose
Population: The analysis population consisted of all participants who received pembrolizumab and contributed blood samples for analysis of Cmax in Part A Cycle 12. There were no participants that contributed data for the analysis of Cmax for the 2 mg/kg arm in Part A of Cycle 12.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Part A: Pembrolizumab 2 mg/kg | Part A: Pembrolizumab 10 mg/kg
Number analyzed (Participants) | 0 | 1
µg/mL |  | 357 (NA) — %CV was not planned to be calculated for ≤2 participants.

11. Secondary Outcome: Maximum Serum Concentration (Cmax) of Pembrolizumab for Cycle 14: Part A
Description: Cmax was the maximum observed concentration of pembrolizumab in serum. Blood sampling was taken for Part A on Day 1 of Cycle 14 at pre-dose and 0-30 minutes post-dose. Cycle 14 length for Part A was 14 days. Cmax is reported as geometric mean with a percent coefficient of variation (%CV). Per protocol, analysis for Cmax in Cycle 14 was only planned for Part A.
Time Frame: Cycle 14 Day 1 pre- and post-dose
Population: The analysis population consisted of all participants who received pembrolizumab and contributed blood samples for analysis of Cmax in Part A Cycle 14. There were no participants that contributed data for the analysis of Cmax for the 2 mg/kg arm in Part A of Cycle 14.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Part A: Pembrolizumab 2 mg/kg | Part A: Pembrolizumab 10 mg/kg
Number analyzed (Participants) | 0 | 1
µg/mL |  | 335 (NA) — %CV was not planned to be calculated for ≤2 participants.

12. Secondary Outcome: Maximum Serum Concentration (Cmax) of Pembrolizumab for Cycle 16: Part A
Description: Cmax was the maximum observed concentration of pembrolizumab in serum. Blood sampling was taken for Part A on Day 1 of Cycle 16 at pre-dose and 0-30 minutes post-dose. Cycle 16 length for Part A was 14 days. Cmax is reported as geometric mean with a percent coefficient of variation (%CV). Per protocol, analysis for Cmax in Cycle 16 was only planned for Part A.
Time Frame: Cycle 16 Day 1 pre- and post-dose
Population: The analysis population consisted of all participants who received pembrolizumab and contributed blood samples for analysis of Cmax in Part A Cycle 16. There were no participants that contributed data for the analysis of Cmax for the 2 mg/kg arm in Part A of Cycle 16.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Part A: Pembrolizumab 2 mg/kg | Part A: Pembrolizumab 10 mg/kg
Number analyzed (Participants) | 0 | 1
µg/mL |  | 348 (NA) — %CV was not planned to be calculated for ≤2 participants.

13. Secondary Outcome: Maximum Serum Concentration (Cmax) of Pembrolizumab for Cycle 18: Part A
Description: Cmax was the maximum observed concentration of pembrolizumab in serum. Blood sampling was taken for Part A on Day 1 of Cycle 18 at pre-dose and 0-30 minutes post-dose. Cycle 18 length for Part A was 14 days. Cmax is reported as geometric mean with a percent coefficient of variation (%CV). Per protocol, analysis for Cmax in Cycle 18 was only planned for Part A.
Time Frame: Cycle 18 Day 1 pre- and post-dose
Population: The analysis population consisted of all participants who received pembrolizumab and contributed blood samples for analysis of Cmax in Part A Cycle 18. There were no participants that contributed data for the analysis of Cmax for the 2 mg/kg arm in Part A of Cycle 18.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Part A: Pembrolizumab 2 mg/kg | Part A: Pembrolizumab 10 mg/kg
Number analyzed (Participants) | 0 | 1
µg/mL |  | 329 (NA) — %CV was not planned to be calculated for ≤2 participants.

14. Secondary Outcome: Time to Maximum Serum Concentration (Tmax) of Pembrolizumab for Cycle 1: Parts A, B, C, D, and E
Description: Tmax was the time required to reach the maximum concentration of pembrolizumab in serum. For Part A, samples were collected on Day 1 at pre-dose, post-dose (to +30 min), 6 hour (hr) (±30 min), and 24hr; Days 2, 3, 8, 15, and 22 (±2 hr for Day 2 to Day 22) after completion of infusion. For Parts B, C, and E, samples were collected on Day 1 at pre-dose, post-dose (to +30 min), and 24hr; Day 5 (96hr was preferred, 72hr or 120hr were also acceptable, ±2 hr), and Day 15 (±24 hr) after completion of infusion. For Part D, samples were collected on Day 1 at pre-dose, post-dose (to +30 min), and 24hr; Day 5 (96hr was preferred, 72hr or 120hr were also acceptable, ±2 hr), Day 15, and Day 22 (±24 hr) after completion of infusion. Cycle 1 length for Part A was 28 days. Cycle 1 length for Parts B, C, and E was 21 days. Cycle 1 length for Part D was 42 days. Tmax is reported as median and full range. Per protocol, analysis for Tmax in Cycle 1 was planned for Parts A, B, C, D, and E.
Time Frame: At designated timepoints in Cycle 1 for Parts A, B, C, D, and E (up to approximately 22 days)
Population: The analysis population consisted of all participants who received pembrolizumab and contributed blood samples for analysis of Tmax in Parts A, B, C, D, and E Cycle 1.
Measure: Median (Full Range); unit: days
Arm/Group | Part A: Pembrolizumab 2 mg/kg | Part A: Pembrolizumab 10 mg/kg | Part B: Pembrolizumab+Cisplatin/Pemetrexed | Part B: Pembrolizumab+Carboplatin/Pemetrexed | Part C: Pembrolizumab+Carboplatin/Paclitaxel | Part C: Pembrolizumab+Carboplatin/Nab-paclitaxel | Part D: Pembrolizumab+Ipilimumab | Part E: Pembrolizumab+Cisplatin/Etoposide | Part E: Pembrolizumab+Carboplatin/Etoposide | Part E: Pembrolizumab+Cisplatin/Etoposide+G-CSF
Number analyzed (Participants) | 3 | 7 | 6 | 6 | 8 | 6 | 6 | 6 | 6 | 3
days | 0.223 [0.00208 to 0.233] | 0.00903 [0.000694 to 0.232] | 1.98 [0.94 to 4.94] | 2.52 [0.033 to 13.91] | 0.028 [0.025 to 1.08] | 0.027 [0.022 to 1.02] | 0.026 [0.024 to 0.029] | 0.026 [0.026 to 0.029] | 0.028 [0.023 to 0.041] | 0.031 [0.025 to 0.033]

15. Secondary Outcome: Time to Maximum Serum Concentration (Tmax) of Pembrolizumab for Cycle 4: Part D
Description: Tmax was the time required to reach the maximum concentration of pembrolizumab in serum. Blood sampling was taken for Part D on Day 22 of Cycle 4 at pre-dose (Day 1 of the following cycle prior to pembrolizumab infusion) and 0-30 minutes post-dose. Cycle length for Part D was 42 days. Tmax is reported as median and full range. Per protocol, analysis for Tmax in Cycle 4 was only planned for Part D.
Time Frame: Cycle 4 Day 22 pre-dose (Day 1 of the following cycle prior to pembrolizumab infusion) and post-dose
Population: The analysis population consisted of all participants who received pembrolizumab and contributed blood samples for Tmax in the Cycle 4 analysis of Part D.
Measure: Median (Full Range); unit: days
Arm/Group | Part D: Pembrolizumab+Ipilimumab
Number analyzed (Participants) | 3
days | 0.026 [0.025 to 0.030]

16. Secondary Outcome: Time to Maximum Serum Concentration (Tmax) of Pembrolizumab for Cycle 8: Parts B, C, and E
Description: Tmax was the time required to reach the maximum concentration of pembrolizumab in serum. Blood sampling was taken for Parts B, C, and E on Day 1 of Cycle 8 at pre-dose and 0-30 minutes post-dose. Cycle 8 for Parts B, C, and E was 21 days. Tmax is reported as median and full range. Per protocol, analysis for Tmax in Cycle 8was planned for Parts B, C, and E.
Time Frame: Cycle 8 Day 1 pre- and post-dose
Population: The analysis population consisted of all participants who received pembrolizumab and contributed blood samples for analysis of Tmax in Parts B, C, and E Cycle 8. There were no participants that contributed data available for the analysis of Tmax for the Pembrolizumab+Cisplatin/Etoposide+G-CSF arm in Part E of Cycle 8.
Measure: Median (Full Range); unit: days
Arm/Group | Part B: Pembrolizumab+Cisplatin/Pemetrexed | Part B: Pembrolizumab+Carboplatin/Pemetrexed | Part C: Pembrolizumab+Carboplatin/Paclitaxel | Part C: Pembrolizumab+Carboplatin/Nab-paclitaxel | Part E: Pembrolizumab+Cisplatin/Etoposide | Part E: Pembrolizumab+Carboplatin/Etoposide | Part E: Pembrolizumab+Cisplatin/Etoposide+G-CSF
Number analyzed (Participants) | 2 | 3 | 1 | 2 | 1 | 3 | 0
days | 0.024 [0.022 to 0.025] | 0.026 [0.025 to 0.026] | 0.028 [0.028 to 0.028] | 0.027 [0.024 to 0.029] | 0.029 [0.029 to 0.029] | 0.026 [0.023 to 0.031] |

17. Secondary Outcome: Trough Concentration (Ctrough) of Pembrolizumab for Cycle 1: Parts A, B, C, D, and E
Description: Ctrough was the lowest concentration of pembrolizumab in serum just before the next dose. Blood sampling for Cycle 1 Ctrough was taken for Parts A, B, C, D, and E on Day 1 of Cycle 2 at pre-dose (prior to Cycle 2 infusion). Cycle 1 length for Part A was 28 days. Cycle 1 length for Parts B, C, and E was 21 days. Cycle 1 length for Part D was 42 days. Ctrough is reported as geometric mean with a percent coefficient of variation (%CV). Per protocol, analysis for Cycle 1 Ctrough was planned for Parts A, B, C, D, and E.
Time Frame: Cycle 2 Day 1 pre-dose
Population: The analysis population consisted of all participants who received pembrolizumab and contributed blood samples for analysis of Cycle 1 Ctrough in Parts A, B, C, D, and E.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Part A: Pembrolizumab 2 mg/kg | Part A: Pembrolizumab 10 mg/kg | Part B: Pembrolizumab+Cisplatin/Pemetrexed | Part B: Pembrolizumab+Carboplatin/Pemetrexed | Part C: Pembrolizumab+Carboplatin/Paclitaxel | Part C: Pembrolizumab+Carboplatin/Nab-paclitaxel | Part D: Pembrolizumab+Ipilimumab | Part E: Pembrolizumab+Cisplatin/Etoposide | Part E: Pembrolizumab+Carboplatin/Etoposide | Part E: Pembrolizumab+Cisplatin/Etoposide+G-CSF
Number analyzed (Participants) | 3 | 6 | 6 | 6 | 6 | 6 | 3 | 5 | 6 | 3
µg/mL | 11.2 (51) | 47.9 (50) | 19.88 (46.61) | 15.79 (33.24) | 9.45 (31.31) | 10.96 (17.19) | 8.26 (16.20) | 14.57 (10.56) | 15.30 (19.82) | 17.88 (9.58)

18. Secondary Outcome: Trough Concentration (Ctrough) of Pembrolizumab for Cycle 2: Part D
Description: Ctrough was the lowest concentration of pembrolizumab in serum just before the next dose. Blood sampling for Cycle 2 Ctrough was taken for Part D on Day 22 of Cycle 2 at pre-dose (prior to Cycle 3 infusion). Cycle 2 length for Part D was 42 days. Ctrough is reported as geometric mean with a percent coefficient of variation (%CV). Per protocol, analysis for Cycle 2 Ctrough was only planned for Part D.
Time Frame: Cycle 2 Day 22 pre-dose
Population: The analysis population consisted of all participants who received pembrolizumab and contributed blood samples for analysis of Cycle 2 Ctrough in Part D.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Part D: Pembrolizumab+Ipilimumab
Number analyzed (Participants) | 5
µg/mL | 20.10 (24.59)

19. Secondary Outcome: Trough Concentration (Ctrough) of Pembrolizumab for Cycle 3: Part D
Description: Ctrough was the lowest concentration of pembrolizumab in serum just before the next dose. Blood sampling for Cycle 3 Ctrough was taken for Part D on Day 22 of Cycle 3 at pre-dose (prior to Cycle 4 infusion). Cycle 3 length for Part D was 42 days. Ctrough is reported as geometric mean with a percent coefficient of variation (%CV).
Time Frame: Cycle 3 Day 22 pre-dose
Population: The analysis population consisted of all participants who received pembrolizumab and contributed blood samples for analysis of Cycle 3 Ctrough in Part D.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Part D: Pembrolizumab+Ipilimumab
Number analyzed (Participants) | 4
µg/mL | 30.30 (19.38)

20. Secondary Outcome: Trough Concentration (Ctrough) of Pembrolizumab for Cycle 3: Parts A, B, C, and E
Description: Ctrough was the lowest concentration of pembrolizumab in serum just before the next dose. Blood sampling for Cycle 3 Ctrough was taken for Parts A, B, C, and E on Day 1 of Cycle 4 at pre-dose (prior to Cycle 4 infusion). Cycle 3 length for Part A was 14 days. Cycle 3 length for Parts B, C, and E was 21 days. Ctrough is reported as geometric mean with a percent coefficient of variation (%CV).
Time Frame: Cycle 4 Day 1 at Pre-dose
Population: The analysis population consisted of all participants who received pembrolizumab and contributed blood samples for analysis of Cycle 3 Ctrough in Parts A, B, C, and E.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Part A: Pembrolizumab 2 mg/kg | Part A: Pembrolizumab 10 mg/kg | Part B: Pembrolizumab+Cisplatin/Pemetrexed | Part B: Pembrolizumab+Carboplatin/Pemetrexed | Part C: Pembrolizumab+Carboplatin/Paclitaxel | Part C: Pembrolizumab+Carboplatin/Nab-paclitaxel | Part E: Pembrolizumab+Cisplatin/Etoposide | Part E: Pembrolizumab+Carboplatin/Etoposide | Part E: Pembrolizumab+Cisplatin/Etoposide+G-CSF
Number analyzed (Participants) | 2 | 4 | 5 | 4 | 3 | 4 | 4 | 5 | 3
µg/mL | 37.2 (13) | 83.0 (265) | 32.71 (30.35) | 25.38 (22.12) | 24.80 (9.28) | 23.63 (4.79) | 32.20 (21.52) | 30.43 (25.67) | 34.31 (22.05)

21. Secondary Outcome: Trough Concentration (Ctrough) of Pembrolizumab for Cycle 4: Part D
Description: Ctrough was the lowest concentration of pembrolizumab in serum just before the next dose. Blood sampling for Cycle 4 Ctrough was taken for Part D on Day 22 of Cycle 4 at pre-dose (prior to Cycle 5 infusion). Cycle 4 length for Part D was 42 days. Ctrough is reported as geometric mean with a percent coefficient of variation (%CV). Per protocol, analysis for Cycle 4 Ctrough was only planned for Part D.
Time Frame: Cycle 4 Day 22 pre-dose
Population: The analysis population consisted of all participants who received pembrolizumab and contributed blood samples for analysis of Cycle 4 Ctrough in Part D.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Part D: Pembrolizumab+Ipilimumab
Number analyzed (Participants) | 4
µg/mL | 28.08 (23.62)

22. Secondary Outcome: Trough Concentration (Ctrough) of Pembrolizumab for Cycle 5: Parts A, B, C, and E
Description: Ctrough was the lowest concentration of pembrolizumab in serum just before the next dose. Blood sampling for Cycle 5 Ctrough was taken for Parts A, B, C, and E on Day 1 of Cycle 6 at pre-dose (prior to Cycle 6 infusion). Cycle 5 length for Part A was 14 days. Cycle 5 length for Parts B, C, and E was 21 days. Ctrough is reported as geometric mean with a percent coefficient of variation (%CV). Per protocol, analysis for Cycle 5 Ctrough was only planned for Parts A, B, C, and E.
Time Frame: Cycle 6 Day 1 pre-dose
Population: The analysis population consisted of all participants who received pembrolizumab and contributed blood samples for analysis of Cycle 5 Ctrough in Parts A, B, C, and E.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Part A: Pembrolizumab 2 mg/kg | Part A: Pembrolizumab 10 mg/kg | Part B: Pembrolizumab+Cisplatin/Pemetrexed | Part B: Pembrolizumab+Carboplatin/Pemetrexed | Part C: Pembrolizumab+Carboplatin/Paclitaxel | Part C: Pembrolizumab+Carboplatin/Nab-paclitaxel | Part E: Pembrolizumab+Cisplatin/Etoposide | Part E: Pembrolizumab+Carboplatin/Etoposide | Part E: Pembrolizumab+Cisplatin/Etoposide+G-CSF
Number analyzed (Participants) | 2 | 3 | 4 | 4 | 3 | 4 | 3 | 4 | 2
µg/mL | 46.5 (12) | 38.3 (1640) | 37.70 (7.95) | 23.84 (69.26) | 35.33 (16.60) | 33.91 (14.66) | 47.82 (14.28) | 38.63 (25.56) | 46.47 (NA) — %CV was not planned to be calculated for ≤2 participants.

23. Secondary Outcome: Trough Concentration (Ctrough) of Pembrolizumab for Cycle 6: Part D
Description: Ctrough was the lowest concentration of pembrolizumab in serum just before the next dose. Blood sampling for Cycle 6 Ctrough was taken for Part D on Day 22 of Cycle 6 at pre-dose (prior to Cycle 7 infusion). Cycle 6 length for Part D was 42 days. Ctrough is reported as geometric mean with a percent coefficient of variation (%CV). Per protocol, analysis for Cycle 6 Ctrough was only planned for Part D.
Time Frame: Cycle 6 Day 22 pre-dose
Population: The analysis population consisted of all participants who received pembrolizumab and contributed blood samples for analysis of Cycle 6 Ctrough in Part D.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Part D: Pembrolizumab+Ipilimumab
Number analyzed (Participants) | 1
µg/mL | 40.10 (NA) — %CV was not planned to be calculated for ≤2 participants

24. Secondary Outcome: Trough Concentration (Ctrough) of Pembrolizumab for Cycle 7: Parts A, B, C, and E
Description: Ctrough was the lowest concentration of pembrolizumab in serum just before the next dose. Blood sampling for Cycle 7 Ctrough was taken for Parts A, B, C, and E on Day 1 of Cycle 8 at pre-dose (prior to Cycle 8 infusion). Cycle 7 length for Part A was 14 days. Cycle 7 length for Parts B, C, and E was 21 days. Ctrough is reported as geometric mean with a percent coefficient of variation (%CV). Per protocol, analysis for Cycle 7 Ctrough was only planned for Parts A, B, C, and E.
Time Frame: Cycle 8 Day 1 pre-dose
Population: The analysis population consisted of all participants who received pembrolizumab and contributed blood samples for analysis of Cycle 7 Ctrough in Parts A, B, C, and E.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Part A: Pembrolizumab 2 mg/kg | Part A: Pembrolizumab 10 mg/kg | Part B: Pembrolizumab+Cisplatin/Pemetrexed | Part B: Pembrolizumab+Carboplatin/Pemetrexed | Part C: Pembrolizumab+Carboplatin/Paclitaxel | Part C: Pembrolizumab+Carboplatin/Nab-paclitaxel | Part E: Pembrolizumab+Cisplatin/Etoposide | Part E: Pembrolizumab+Carboplatin/Etoposide | Part E: Pembrolizumab+Cisplatin/Etoposide+G-CSF
Number analyzed (Participants) | 2 | 1 | 2 | 3 | 1 | 4 | 1 | 3 | 1
µg/mL | 54.9 (13) | 134 (NA) — %CV was not planned to be calculated for ≤2 participants | 39.33 (NA) — %CV was not planned to be calculated for ≤2 participants | 37.44 (8.87) | 42.70 (NA) — %CV was not planned to be calculated for ≤2 participants | 32.44 (29.15) | 54.0 (NA) — %CV was not planned to be calculated for ≤2 participants | 48.92 (15.61) | 43.10 (NA) — %CV was not planned to be calculated for ≤2 participants

25. Secondary Outcome: Trough Concentration (Ctrough) of Pembrolizumab for Cycle 8: Part D
Description: Ctrough was the lowest concentration of pembrolizumab in serum just before the next dose. Blood sampling for Cycle 8 Ctrough was taken for Part D on Day 22 of Cycle 8 at pre-dose (prior to Cycle 9 infusion). Cycle 8 length for Part D was 42 days. Ctrough is reported as geometric mean with a percent coefficient of variation (%CV). Per protocol, analysis for Cycle 8 Ctrough was only planned for Part D.
Time Frame: Cycle 8 Day 22 pre-dose
Population: The analysis population consisted of all participants who received pembrolizumab and contributed blood samples for analysis of Cycle 8 Ctrough in Part D.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Part D: Pembrolizumab+Ipilimumab
Number analyzed (Participants) | 1
µg/mL | 35.20 (NA) — %CV was not planned to be calculated for ≤2 participants

26. Secondary Outcome: Trough Concentration (Ctrough) of Pembrolizumab for Cycle 9: Part A
Description: Ctrough was the lowest concentration of pembrolizumab in serum just before the next dose. Blood sampling for Cycle 9 Ctrough was taken for Part A on Day 1 of Cycle 10 at pre-dose (prior to Cycle 10 infusion). Cycle 9 length for Part A was 14 days. Ctrough is reported as geometric mean with a percent coefficient of variation (%CV). Per protocol, analysis for Cycle 9 Ctrough was only planned for Part A.
Time Frame: Cycle 10 Day 1 pre-dose
Population: The analysis population consisted of all participants who received pembrolizumab and contributed blood samples for analysis of Cycle 9 Ctrough in Part A.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Part A: Pembrolizumab 2 mg/kg | Part A: Pembrolizumab 10 mg/kg
Number analyzed (Participants) | 1 | 1
µg/mL | 68.4 (NA) — %CV was not planned to be calculated for ≤2 participants. | 125 (NA) — %CV was not planned to be calculated for ≤2 participants.

27. Secondary Outcome: Trough Concentration (Ctrough) of Pembrolizumab for Cycle 10: Part D
Description: Ctrough was the lowest concentration of pembrolizumab in serum just before the next dose. Blood sampling for Cycle 10 Ctrough was taken for Part D on Day 22 of Cycle 10 at pre-dose (prior to Cycle 11 infusion). Cycle 10 length for Part D was 42 days. Ctrough is reported as geometric mean with a percent coefficient of variation (%CV). Per protocol, analysis for Cycle 10 Ctrough was only planned for Part D.
Time Frame: Cycle 10 Day 22 pre-dose
Population: The analysis population consisted of all participants who received pembrolizumab and contributed blood samples for analysis of Cycle 10 Ctrough in Part D.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Part D: Pembrolizumab+Ipilimumab
Number analyzed (Participants) | 1
µg/mL | 36.30 (NA) — %CV was not planned to be calculated for ≤2 participants

28. Secondary Outcome: Trough Concentration (Ctrough) of Pembrolizumab for Cycle 11: Parts A, B, C, and E
Description: Ctrough was the lowest concentration of pembrolizumab in serum just before the next dose. Blood sampling for Cycle 11 Ctrough was taken for Parts A, B, C, and E on Day 1 of Cycle 12 at pre-dose (prior to Cycle 12 infusion). Cycle 11 length for Part A was 14 days. Cycle 11 length for Parts B, C, and E was 21 days. Ctrough is reported as geometric mean with a percent coefficient of variation (%CV). Per protocol, analysis for Cycle 11 Ctrough was only planned for Parts A, B, C, and E.
Time Frame: Cycle 12 Day 1 Pre-dose
Population: The analysis population consisted of all participants who received pembrolizumab and contributed blood samples for analysis of Cycle 11 Ctrough in Parts A, B, C, and E. There were no participants that contributed data for the analysis of Ctrough for the Part A 2 mg/kg arm and Part E Pembrolizumab+Carboplatin/Etoposide and Pembrolizumab+Cisplatin/Etoposide+G-CSF arms.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Part A: Pembrolizumab 2 mg/kg | Part A: Pembrolizumab 10 mg/kg | Part B: Pembrolizumab+Cisplatin/Pemetrexed | Part B: Pembrolizumab+Carboplatin/Pemetrexed | Part C: Pembrolizumab+Carboplatin/Paclitaxel | Part C: Pembrolizumab+Carboplatin/Nab-paclitaxel | Part E: Pembrolizumab+Cisplatin/Etoposide | Part E: Pembrolizumab+Carboplatin/Etoposide | Part E: Pembrolizumab+Cisplatin/Etoposide+G-CSF
Number analyzed (Participants) | 0 | 1 | 1 | 3 | 1 | 1 | 1 | 0 | 0
µg/mL |  | 159 (NA) — %CV was not planned to be calculated for ≤2 participants. | 39.30 (NA) — %CV was not planned to be calculated for ≤2 participants. | 45.00 (6.84) | 32.60 (NA) — %CV was not planned to be calculated for ≤2 participants. | 57.80 (NA) — %CV was not planned to be calculated for ≤2 participants. | 52.20 (NA) — %CV was not planned to be calculated for ≤2 participants. |  |

29. Secondary Outcome: Trough Concentration (Ctrough) of Pembrolizumab for Cycle 12: Part D
Description: Ctrough was the lowest concentration of pembrolizumab in serum just before the next dose. Blood sampling for Cycle 12 Ctrough was taken for Part D on Day 22 of Cycle 12 at pre-dose (prior to Cycle 13 infusion). Cycle 12 length for Part D was 42 days. Ctrough is reported as geometric mean with a percent coefficient of variation (%CV). Per protocol, analysis for Cycle 12 Ctrough was only planned for Part D.
Time Frame: Cycle 12 Day 22 pre-dose
Population: The analysis population consisted of all participants who received pembrolizumab and contributed blood samples for analysis of Cycle 12 Ctrough in Part D.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Part D: Pembrolizumab+Ipilimumab
Number analyzed (Participants) | 1
µg/mL | 30.90 (NA) — %CV was not planned to be calculated for ≤2 participants

30. Secondary Outcome: Trough Concentration (Ctrough) of Pembrolizumab for Cycle 13: Part A
Description: Ctrough was the lowest concentration of pembrolizumab in serum just before the next dose. Blood sampling for Cycle 13 Ctrough was taken for Part A on Day 1 of Cycle 14 at pre-dose (prior to Cycle 14 infusion). Cycle 13 length for Part A was 14 days. Ctrough is reported as geometric mean with a percent coefficient of variation (%CV). Per protocol, analysis for Cycle 13 Ctrough was only planned for Part A.
Time Frame: Cycle 14 Day 1 pre-dose
Population: The analysis population consisted of all participants who received pembrolizumab and contributed blood samples for analysis of Cycle 13 Ctrough in Part A. There were no participants that contributed data for the analysis of Ctrough for the Part A 2 mg/kg arm.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Part A: Pembrolizumab 2 mg/kg | Part A: Pembrolizumab 10 mg/kg
Number analyzed (Participants) | 0 | 1
µg/mL |  | 147 (NA) — %CV was not planned to be calculated for ≤2 participants.

31. Secondary Outcome: Trough Concentration (Ctrough) of Pembrolizumab for Cycle 14: Part D
Description: Ctrough was the lowest concentration of pembrolizumab in serum just before the next dose. Blood sampling for Cycle 14 Ctrough was taken for Part D on Day 22 of Cycle 14 at pre-dose (prior to Cycle 15 infusion). Cycle 14 length for Part D was 42 days. Ctrough is reported as geometric mean with a percent coefficient of variation (%CV). Per protocol, analysis for Cycle 14 Ctrough was only planned for Part D.
Time Frame: Cycle 14 Day 22 pre-dose
Population: The analysis population consisted of all participants who received pembrolizumab and contributed blood samples for analysis of Cycle 14 Ctrough in Part D.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Part D: Pembrolizumab+Ipilimumab
Number analyzed (Participants) | 1
µg/mL | 28.40 (NA) — %CV was not planned to be calculated for ≤2 participants

32. Secondary Outcome: Trough Concentration (Ctrough) of Pembrolizumab for Cycle 15: Parts A, B, C, and E
Description: Ctrough was the lowest concentration of pembrolizumab in serum just before the next dose. Blood sampling was taken for Parts A, B, C, and E on Day 1 of Cycle 16 at pre-dose (prior to Cycle 16 infusion). Cycle 15 length for Part A was 14 days. Cycle 15 length for Parts B, C, and E was 21 days. Ctrough is reported as geometric mean with a percent coefficient of variation (%CV). Per protocol, analysis for Cycle 15 Ctrough was only planned for Parts A, B, C, and E.
Time Frame: Cycle 16 Day 1 pre-dose
Population: The analysis population consisted of all participants who received pembrolizumab and contributed blood samples for analysis of Cycle 15 Ctrough in Parts A, B, C, and E. There were no participants that contributed data for the analysis of Ctrough for the Part A 2 mg/kg arm; Part C Pembrolizumab+Carboplatin/Paclitaxel and Pembrolizumab+Carboplatin/Nab-paclitaxel arms; and Part E Pembrolizumab+Carboplatin/Etoposide and Pembrolizumab+Cisplatin/Etoposide+G-CSF arms.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Part A: Pembrolizumab 2 mg/kg | Part A: Pembrolizumab 10 mg/kg | Part B: Pembrolizumab+Cisplatin/Pemetrexed | Part B: Pembrolizumab+Carboplatin/Pemetrexed | Part C: Pembrolizumab+Carboplatin/Paclitaxel | Part C: Pembrolizumab+Carboplatin/Nab-paclitaxel | Part E: Pembrolizumab+Cisplatin/Etoposide | Part E: Pembrolizumab+Carboplatin/Etoposide | Part E: Pembrolizumab+Cisplatin/Etoposide+G-CSF
Number analyzed (Participants) | 0 | 1 | 1 | 2 | 0 | 0 | 1 | 0 | 0
µg/mL |  | 199 (NA) — %CV was not planned to be calculated for ≤2 participants. | 47.50 (NA) — %CV was not planned to be calculated for ≤2 participants. | 56.27 (NA) — %CV was not planned to be calculated for ≤2 participants. |  |  | 52.50 (NA) — %CV was not planned to be calculated for ≤2 participants. |  |

33. Secondary Outcome: Trough Concentration (Ctrough) of Pembrolizumab for Cycle 16: Part D
Description: Ctrough was the lowest concentration of pembrolizumab in serum just before the next dose. Blood sampling for Cycle 16 Ctrough was taken for Part D on Day 22 of Cycle 16 at pre-dose (prior to Cycle 17 infusion). Cycle 16 length for Part D was 42 days. Ctrough is reported as geometric mean with a percent coefficient of variation (%CV). Per protocol, analysis for Cycle 16 Ctrough was only planned for Part D.
Time Frame: Cycle 16 Day 22 pre-dose
Population: The analysis population consisted of all participants who received pembrolizumab and contributed blood samples for analysis of Cycle 16 Ctrough in Part D.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Part D: Pembrolizumab+Ipilimumab
Number analyzed (Participants) | 1
µg/mL | 30.70 (NA) — %CV was not planned to be calculated for ≤2 participants

34. Secondary Outcome: Trough Concentration (Ctrough) of Pembrolizumab for Cycle 17: Part A
Description: Ctrough was the lowest concentration of pembrolizumab in serum just before the next dose. Blood sampling was taken for Part A on Day 1 of Cycle 18 at pre-dose (prior to Cycle 18 infusion). Cycle 17 length for Part A was 14 days. Ctrough is reported as geometric mean with a percent coefficient of variation (%CV). Per protocol, analysis for Cycle 17 Ctrough was planned for Part A.
Time Frame: Cycle 18 Day 1 pre-dose
Population: The analysis population consisted of all participants who received pembrolizumab and contributed blood samples for analysis of Cycle 17 Ctrough in Part A. There were no participants that contributed data for the analysis of Ctrough for the Part A 2 mg/kg arm.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Part A: Pembrolizumab 2 mg/kg | Part A: Pembrolizumab 10 mg/kg
Number analyzed (Participants) | 0 | 1
µg/mL |  | 125 (NA) — %CV cannot be calculated for 1 participant.

35. Secondary Outcome: Trough Concentration (Ctrough) of Pembrolizumab for Cycle 19: Parts B, C, and E
Description: Ctrough was the lowest concentration of pembrolizumab in serum just before the next dose. Blood sampling was taken for Parts B, C, and E on Day 1 of Cycle 20 at pre-dose (prior to Cycle 20 infusion). Cycle 19 length for Parts B, C, and E was 21 days. Ctrough is reported as geometric mean with a percent coefficient of variation (%CV). Per protocol, analysis for Cycle 19 Ctrough was only planned for Parts B, C, and E.
Time Frame: Cycle 20 Day 1 Pre-dose
Population: The analysis population consisted of all participants who received pembrolizumab and contributed blood samples for analysis of Cycle 19 Ctrough in Parts B, C, and E. There were no participants that contributed data for the analysis of Ctrough for the Part C Pembrolizumab+Carboplatin/Paclitaxel and Pembrolizumab+Carboplatin/Nab-paclitaxel arms; and Part E Pembrolizumab+Cisplatin/Etoposide, Pembrolizumab+Carboplatin/Etoposide, and Pembrolizumab+Cisplatin/Etoposide+G-CSF arms.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Part B: Pembrolizumab+Cisplatin/Pemetrexed | Part B: Pembrolizumab+Carboplatin/Pemetrexed | Part C: Pembrolizumab+Carboplatin/Paclitaxel | Part C: Pembrolizumab+Carboplatin/Nab-paclitaxel | Part E: Pembrolizumab+Cisplatin/Etoposide | Part E: Pembrolizumab+Carboplatin/Etoposide | Part E: Pembrolizumab+Cisplatin/Etoposide+G-CSF
Number analyzed (Participants) | 1 | 2 | 0 | 0 | 0 | 0 | 0
µg/mL | 48.50 (NA) — %CV was not planned to be calculated for ≤2 participants. | 50.98 (NA) — %CV was not planned to be calculated for ≤2 participants. |  |  |  |  |

36. Secondary Outcome: Trough Concentration (Ctrough) of Pembrolizumab for Cycle 23: Parts B, C, and E
Description: Ctrough was the lowest concentration of pembrolizumab in serum just before the next dose. Blood sampling was taken for Parts B, C, and E on Day 1 of Cycle 24 at pre-dose (prior to Cycle 24 infusion). Cycle 23 length for Parts B, C, and E was 21 days. Ctrough is reported as geometric mean with a percent coefficient of variation (%CV). Per protocol, analysis for Cycle 23 Ctrough was only planned for Parts B, C, and E.
Time Frame: Cycle 24 Day 1 Pre-dose
Population: The analysis population consisted of all participants who received pembrolizumab and contributed blood samples for analysis of Cycle 23 Ctrough in Parts B, C, and E. There were no participants that contributed data for the analysis of Ctrough for the Part C Pembrolizumab+Carboplatin/Paclitaxel and Pembrolizumab+Carboplatin/Nab-paclitaxel arms; and Part E Pembrolizumab+Cisplatin/Etoposide, Pembrolizumab+Carboplatin/Etoposide, and Pembrolizumab+Cisplatin/Etoposide+G-CSF arms.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Part B: Pembrolizumab+Cisplatin/Pemetrexed | Part B: Pembrolizumab+Carboplatin/Pemetrexed | Part C: Pembrolizumab+Carboplatin/Paclitaxel | Part C: Pembrolizumab+Carboplatin/Nab-paclitaxel | Part E: Pembrolizumab+Cisplatin/Etoposide | Part E: Pembrolizumab+Carboplatin/Etoposide | Part E: Pembrolizumab+Cisplatin/Etoposide+G-CSF
Number analyzed (Participants) | 1 | 2 | 0 | 0 | 0 | 0 | 0
µg/mL | 42.40 (NA) — %CV was not planned to be calculated for ≤2 participants. | 51.72 (NA) — %CV was not planned to be calculated for ≤2 participants. |  |  |  |  |

37. Secondary Outcome: Trough Concentration (Ctrough) of Pembrolizumab for Cycle 27: Parts B, C, and E
Description: Ctrough was the lowest concentration of pembrolizumab in serum just before the next dose. Blood sampling was taken for Parts B, C, and E on Day 1 of Cycle 28 at pre-dose (prior to Cycle 28 infusion). Cycle 27 length for Parts B, C, and E was 21 days. Ctrough is reported as geometric mean with a percent coefficient of variation (%CV). Per protocol, analysis for Cycle 27 Ctrough was only planned for Parts B, C, and E.
Time Frame: Cycle 28 Day 1 Pre-dose
Population: The analysis population consisted of all participants who received pembrolizumab and contributed blood samples for analysis of Cycle 27 Ctrough in Parts B, C, and E. There were no participants that contributed data for the analysis of Ctrough for the Part C Pembrolizumab+Carboplatin/Paclitaxel and Pembrolizumab+Carboplatin/Nab-paclitaxel arms; and Part E Pembrolizumab+Cisplatin/Etoposide, Pembrolizumab+Carboplatin/Etoposide, and Pembrolizumab+Cisplatin/Etoposide+G-CSF arms.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Part B: Pembrolizumab+Cisplatin/Pemetrexed | Part B: Pembrolizumab+Carboplatin/Pemetrexed | Part C: Pembrolizumab+Carboplatin/Paclitaxel | Part C: Pembrolizumab+Carboplatin/Nab-paclitaxel | Part E: Pembrolizumab+Cisplatin/Etoposide | Part E: Pembrolizumab+Carboplatin/Etoposide | Part E: Pembrolizumab+Cisplatin/Etoposide+G-CSF
Number analyzed (Participants) | 1 | 1 | 0 | 0 | 0 | 0 | 0
µg/mL | 53.90 (NA) — %CV was not planned to be calculated for ≤2 participants. | 68.20 (NA) — %CV was not planned to be calculated for ≤2 participants. |  |  |  |  |

38. Secondary Outcome: Area Under the Concentration Time Curve From 0-28 Days (AUC 0-28) for Part A Cycle 1
Description: AUC 0-28 was the AUC of pembrolizumab from time zero to 28 days after dosing. Blood sampling was taken at the following timepoints: Part A Cycle 1 Day 1 at pre-dose, 0-30 minutes post-dose, and at 6, 24, 48, 168, 336, 504 hours after completion of pembrolizumab infusion and Day 1 of Cycle 2 pre-dose. Cycle 1 length was 28 days. AUC 0-28 is reported as geometric mean with a percent coefficient of variation. Per protocol, analysis for AUC 0-28 was only planned for Part A Cycle 1.
Time Frame: At designated timepoints in Cycle 1 for Part A (Up to approximately 28 days)
Population: The analysis population consisted of all participants who received pembrolizumab and had blood samples assessed for AUC 0-28 in Part A Cycle 1.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg•day/mL
Arm/Group | Part A: Pembrolizumab 2 mg/kg | Part A: Pembrolizumab 10 mg/kg
Number analyzed (Participants) | 3 | 7
µg•day/mL | 507 (20) | 2219 (32)

39. Secondary Outcome: Area Under the Concentration Time Curve From 0-Infinity (AUC 0-inf) for Part A Cycle 1
Description: AUC 0-inf was the AUC of pembrolizumab from time zero to infinity after dosing. Blood sampling was taken at the following timepoints: Part A Cycle 1 Day 1 at pre-dose, 0-30 minutes post-dose, and at 6, 24, 48, 168, 336, 504 hours after completion of pembrolizumab infusion and Day 1 of Cycle 2 pre-dose. Cycle 1 length was 28 days. AUC 0-inf is reported as geometric mean with a percent coefficient of variation. Per protocol, analysis for AUC 0-inf was only planned for Part A Cycle 1.
Time Frame: At designated timepoints in Cycle 1 for Part A (Up to approximately 28 days)
Population: The analysis population consisted of all participants who received pembrolizumab and had blood samples assessed for AUC 0-inf in Part A Cycle 1.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg•day/mL
Arm/Group | Part A: Pembrolizumab 2 mg/kg | Part A: Pembrolizumab 10 mg/kg
Number analyzed (Participants) | 3 | 7
µg•day/mL | 812 (45) | 3410 (56)

40. Secondary Outcome: Terminal Half-Life (t1/2) of Pembrolizumab Over Time for Part A Cycle 1
Description: t1/2 was the time required to divide the pembrolizumab concentration by two after reaching pseudo-equilibrium. Blood sampling was taken at the following timepoints: Part A Cycle 1 Day 1 at pre-dose, 0-30 minutes post-dose, and at 6, 24, 48, 168, 336, 504 hours after completion of pembrolizumab infusion and pre-dose Day 1 of the following cycle prior to pembrolizumab infusion. Cycle 1 length A was 28 days. t1/2 is reported as geometric mean with a percent coefficient of variation. Per protocol, analysis for t1/2 was only planned for Part A Cycle 1.
Time Frame: At designated timepoints in Cycle 1 for Part A (Up to approximately 28 days)
Population: The analysis population consisted of all participants who received pembrolizumab and had blood samples assessed for t1/2 in Part A Cycle 1.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: days
Arm/Group | Part A: Pembrolizumab 2 mg/kg | Part A: Pembrolizumab 10 mg/kg
Number analyzed (Participants) | 3 | 7
days | 18.4 (56) | 18.1 (68)

41. Secondary Outcome: Volume of Distribution (Vz) of Pembrolizumab Over Time for Part A Cycle 1
Description: Vz was the volume of distribution during the terminal phase. Blood sampling was taken at the following timepoints: Part A Cycle 1 Day 1 at pre-dose, 0-30 minutes post-dose, and at 6, 24, 48, 168, 336, 504 hours after completion of pembrolizumab infusion and Day 1 of Cycle 2 prior to pembrolizumab infusion. Cycle 1 length A was 28 days. Vz is reported as geometric mean with a percent coefficient of variation. Per protocol, analysis for Vz was only planned for Part A Cycle 1.
Time Frame: At designated timepoints in Cycle 1 for Part A (Up to approximately 28 days)
Population: The analysis population consisted of all participants who received pembrolizumab and had blood samples assessed for Vz in Part A Cycle 1.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/kg
Arm/Group | Part A: Pembrolizumab 2 mg/kg | Part A: Pembrolizumab 10 mg/kg
Number analyzed (Participants) | 3 | 7
mL/kg | 65.3 (21) | 76.5 (34)

42. Secondary Outcome: Clearance (CL) of Pembrolizumab Over Time for Part A Cycle 1
Description: CL was the volume of plasma from which pembrolizumab was eliminated per unit time. Blood sampling was taken at the following timepoints: Part A Cycle 1 Day 1 at pre-dose, 0-30 minutes post-dose, and at 6, 24, 48, 168, 336, 504 hours after completion of pembrolizumab infusion and Day 1 of Cycle 2 prior to pembrolizumab infusion. Cycle 1 length A was 28 days. CL is reported as geometric mean with a percent coefficient of variation. Per protocol, analysis for CL was only planned for Part A Cycle 1.
Time Frame: At designated timepoints in Cycle 1 for Part A (Up to approximately 28 days)
Population: The analysis population consisted of all participants who received pembrolizumab and had blood samples assessed for CL in Part A Cycle 1.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/day/kg
Arm/Group | Part A: Pembrolizumab 2 mg/kg | Part A: Pembrolizumab 10 mg/kg
Number analyzed (Participants) | 3 | 7
mL/day/kg | 2.46 (45) | 2.93 (56)

ADVERSE EVENTS:
Time Frame: Up to approximately 51.3 months
Description: Serious and Non-serious AEs presented for participants who received ≥1 dose of study drug. Per protocol, MedDRA preferred terms "Neoplasm progression (NP)", "Malignant NP" & "Disease progression" not related to study treatment are excluded as AEs. Data for all-cause mortality presented for randomized participants.
Arm/Group | Part A: Pembrolizumab 2 mg/kg | Part A: Pembrolizumab 10 mg/kg | Part B: Pembrolizumab+Cisplatin/Pemetrexed | Part B: Pembrolizumab+Carboplatin/Pemetrexed | Part C: Pembrolizumab+Carboplatin/Paclitaxel | Part C: Pembrolizumab+Carboplatin/Nabpaclitaxel | Part D: Pembrolizumab+Ipilimumab | Part E: Pembrolizumab+Cisplatin/Etoposide | Part E: Pembrolizumab+Carboplatin/Etoposide | Part E: Pembrolizumab+Cisplatin/Etoposide+G-CSF
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/7 | 5/6 | 5/6 | 5/8 | 3/6 | 4/6 | 5/6 | 5/6 | 2/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/7 | 2/6 | 5/6 | 3/8 | 3/6 | 1/6 | 3/6 | 2/6 | 0/3
Other Adverse Events (participants affected / at risk) | 3/3 | 7/7 | 6/6 | 6/6 | 8/8 | 6/6 | 5/6 | 6/6 | 6/6 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Pembrolizumab 2 mg/kg (N=3) | Part A: Pembrolizumab 10 mg/kg (N=7) | Part B: Pembrolizumab+Cisplatin/Pemetrexed (N=6) | Part B: Pembrolizumab+Carboplatin/Pemetrexed (N=6) | Part C: Pembrolizumab+Carboplatin/Paclitaxel (N=8) | Part C: Pembrolizumab+Carboplatin/Nabpaclitaxel (N=6) | Part D: Pembrolizumab+Ipilimumab (N=6) | Part E: Pembrolizumab+Cisplatin/Etoposide (N=6) | Part E: Pembrolizumab+Carboplatin/Etoposide (N=6) | Part E: Pembrolizumab+Cisplatin/Etoposide+G-CSF (N=3)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Laryngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lichenoid keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Pembrolizumab 2 mg/kg (N=3) | Part A: Pembrolizumab 10 mg/kg (N=7) | Part B: Pembrolizumab+Cisplatin/Pemetrexed (N=6) | Part B: Pembrolizumab+Carboplatin/Pemetrexed (N=6) | Part C: Pembrolizumab+Carboplatin/Paclitaxel (N=8) | Part C: Pembrolizumab+Carboplatin/Nabpaclitaxel (N=6) | Part D: Pembrolizumab+Ipilimumab (N=6) | Part E: Pembrolizumab+Cisplatin/Etoposide (N=6) | Part E: Pembrolizumab+Carboplatin/Etoposide (N=6) | Part E: Pembrolizumab+Cisplatin/Etoposide+G-CSF (N=3)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 4 (5) | 4 (7) | 3 (3) | 6 (10) | 1 (1) | 2 (3) | 6 (6) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 4 (10) | 4 (10) | 4 (8) | 6 (16) | 0 (0) | 6 (12) | 6 (10) | 2 (4)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 1 (6) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 5 (11) | 2 (8) | 5 (9) | 6 (20) | 0 (0) | 5 (12) | 6 (10) | 2 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (3) | 2 (6) | 2 (8) | 2 (2) | 4 (9) | 0 (0) | 1 (1) | 2 (4) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uveitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angular cheilitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (2) | 0 (0) | 4 (9) | 3 (3) | 4 (6) | 3 (3) | 1 (1) | 6 (8) | 3 (3) | 3 (4)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (2) | 1 (4) | 6 (20) | 5 (5) | 3 (5) | 5 (7) | 0 (0) | 3 (5) | 2 (3) | 3 (3)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Proctitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (4) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 2 (4) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Extravasation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Face oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (2) | 3 (3) | 1 (6) | 1 (1) | 1 (4) | 1 (1) | 1 (1) | 1 (3) | 0 (0) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion site extravasation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 1 (1) | 1 (1) | 4 (4) | 3 (5) | 4 (4) | 3 (5) | 3 (3) | 0 (0) | 2 (2) | 1 (1)
Oedema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 3 (5) | 2 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (4)
Pyrexia (General disorders) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 3 (6) | 2 (2) | 3 (4) | 1 (1) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatotoxicity (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contrast media allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Clostridial infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (3) | 1 (2) | 0 (0) | 1 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Parotitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinea pedis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 3 (3) | 2 (2) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 1 (1)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood cholesterol increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood thyroid stimulating hormone decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
QRS axis abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 6 (14) | 3 (4) | 4 (6) | 6 (9) | 2 (2) | 3 (6) | 5 (5) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (2) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 3 (4) | 2 (2) | 1 (3) | 2 (3) | 2 (4) | 0 (0) | 2 (4) | 1 (1) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypersomnia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 5 (5) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Restlessness (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 4 (5) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 1 (3) | 1 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 5 (5) | 5 (5) | 0 (0) | 3 (3) | 2 (2) | 2 (2)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palmoplantar pustulosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 3 (3) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (2) | 1 (1) | 3 (6) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vasculitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-24): https://cdn.clinicaltrials.gov/large-docs/79/NCT01840579/Prot_SAP_000.pdf